CLINICAL TRIAL: NCT02381314
Title: A Phase 1, Open-Label, Dose Escalation Study of MGA271 in Combination With Ipilimumab in Patients With Melanoma, Non-Small Cell Lung Cancer, and Other Cancers
Brief Title: Safety Study of Enoblituzumab (MGA271) in Combination With Ipilimumab in Refractory Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGA271-02
Record Dates: First submitted 2015-02-20; First posted 2015-03-06 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Melanoma; Non Small Cell Lung Cancer
Keywords: Other B7-H3 expressing cancers
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- enoblituzumab plus ipilimumab (Experimental): Enoblituzumab: Fc-optimized, humanized monoclonal antibody. Ipilimumab: Yervoy; recombinant, fully humanized IgG-1 CTLA-4 blocking antibody approved by the US Food and Drug Administration and the European Medicines Agency for the treatment of unresectable or metastatic melanoma.
  Interventions: Biological: enoblituzumab plus ipilimumab

INTERVENTIONS:
Biological: enoblituzumab plus ipilimumab — enoblituzumab is administered by IV infusion once per week. Ipilimumab is administered by IV infusion every 3 weeks for up to 4 doses.
  Other Names: enoblituzumab (MGA271); ipilimumab (Yervoy)

SUMMARY:
The purpose of this study is to evaluate the safety of enoblituzumab (MGA271) in combination with Yervoy (ipilimumab) when given to patients with B7-H3-expressing melanoma, squamous cell carcinoma of the head and neck (SCCHN), non small cell lung cancer (NSCLC) and other B7-H3 expressing cancers. The study will also evaluate what is the best dose of enoblituzumab to use when given with ipilimumab. Assessments will also be done to see how the drug acts in the body (pharmacokinetics (PK), pharmacodynamics) and to evaluate potential anti-tumor activity of enoblituzumab in combination with ipilimumab.

DETAILED DESCRIPTION:
This study is a Phase 1 open-label, dose escalation, and cohort expansion study of enoblituzumab administered intravenously (IV) on a weekly schedule for up to 51 doses in combination with IV ipilimumab administered on an every-3-week schedule for 4 doses.

The dose escalation phase is designed to characterize the safety and tolerability of the combination of enoblituzumab and ipilimumab and to define the maximum tolerated or administered dose (MTD/MAD) in patients with B7-H3 expressing mesothelioma, urothelial cancer, NSCLC, SCCHN, Clear cell renal cell carcinoma (ccRCC), ovarian cancer, melanoma, thyroid cancer, Triple negative breast cancer (TNBC), pancreatic cancer, colon cancer, soft tissue sarcoma, or prostate cancer.

The cohort expansion phase, 2 cohorts of 16 patients each will be enrolled to further evaluate the safety and potential efficacy of the combination administered at the MTD/MAD dose in patients with melanoma and NSCLC.

All tumor evaluations will be carried out by both Response Evaluation Criteria in Solid Tumors (RECIST) and immune-related response criteria (irRC).

ELIGIBILITY:
Inclusion Criteria - Cohort Expansion Phase:

* Histologically-proven, unresectable, locally advanced or metastatic melanoma or NSCLC

  * Melanoma: Advanced or metastatic melanoma patients may be systemic therapy naïve or may have received systemic treatment for unresectable locally advanced or metastatic disease. A patient who previously received systemic therapy must have had progression on a checkpoint inhibitor (e.g., anti-PD-L1, anti-PD-1, anti-CTLA-4) as the most recent prior therapy.
  * NSCLC: NSCLC that has progressed during or following 1 or more prior systemic therapies for unresectable locally advanced or metastatic disease. Patients who are intolerant of, or have refused treatment with standard first line cancer therapy, will be allowed to enroll. Patients must not have had more than 5 prior systemic regimens (excluding experimental therapies) for unresectable locally advanced or metastatic disease.
* B7-H3 expression is not required for eligibility in this study; however, tumor expression of B7-H3 will be evaluated for all patients.
* Measurable disease per RECIST 1.1 criteria
* ECOG performance status 0 or 1
* Acceptable laboratory parameters and adequate organ reserve.

Exclusion Criteria - Cohort Expansion Phase:

* Patients with a history of symptomatic central nervous system metastases, unless treated and asymptomatic
* Patients with history of autoimmune disease with certain exceptions
* History of allogeneic bone marrow, stem cell, or solid organ transplant
* Treatment with systemic cancer therapy or investigational therapy within 4 weeks; radiation within 2 weeks; trauma or major surgery within 4 weeks
* History of clinically-significant cardiovascular disease; gastrointestinal perforation; gastrointestinal bleeding, acute pancreatitis or diverticulitis within 4 weeks;
* Active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 7 days; positive for human immunodeficiency virus or AIDS, hepatitis B or C.
* Known hypersensitivity to recombinant proteins, polysorbate 80, or any excipient contained in the drug or vehicle formulation for MGA271 or ipilimumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 1 year
  Adverse events, serious adverse events

SECONDARY OUTCOMES:
Peak plasma concentration | 7 weeks
  PK of MGA271 in combination with ipilimumab
Number of participants that develop anti-drug antibodies | 7 weeks
  Proportion of patients who develop anti-MGA271 antibodies, immunogenicity
Change in tumor volume | Weeks 9, 18, 27, 39, and 51
  Anti-tumor activity of MGA271 in combination with ipilimumab using both conventional RECIST 1.1 and immune-related RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — MacroGenics
Locations (10):
- United States (10):
  - UCLA Hematology-Oncology Clinic, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Chicago, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Center for Oncology and Blood Disorders, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided